CLINICAL TRIAL: NCT03146195
Title: The 3D Reconstruction Research of Pelvic Organ Prolapse Disease and the Establishment of Assessment for Space Coordinates
Brief Title: The 3D Reconstruction Research of Pelvic Organ Prolapse Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC2013032-3
Record Dates: First submitted 2017-03-28; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2016-09

CONDITIONS: Pelvic Organ Prolapse; Normal Pelvic Floor
Keywords: pelvic organ prolapse; dynamic magnetic resonance imaging; three-dimensional reconstruction; space coordinates
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- POP: Female patients with pelvic organ prolapse,such as: cystocele, uterine prolapse, the vault prolapse, rectal prolapse ,undergo pelvic floor reconstruction surgery.Before and after sugery,take dynamic magnetic resonance imaging scan.
  Interventions: Other: Dynamic Magnetic resonance imaging
- Non-POP: Females with normal pelvic floor support,don't need pelvic floor reconstruction surgery,only take once dynamic magnetic resonance imaging scan.
  Interventions: Other: Dynamic Magnetic resonance imaging

INTERVENTIONS:
Other: Dynamic Magnetic resonance imaging

SUMMARY:
Female pelvic organ prolapse (FPOP) is one of the main diseases affecting the quality of life of middle aged and elderly women in non-neoplastic diseases. An aging population makes the incidence of this disease to increase year by year. Surgical operation is the main treatment. While the recurrence rate of classic repair surgery is high, the method of patch implantation reinforces the supporting force, which significantly reduce the recurrence rate. However, this method is costly and is associated with complications which may trigger new symptoms. As such, there is still no perfect surgical method. The main reason for this is that the assessment method of pelvic defects is crude and indirect, which results in the diagnosis of FPOP only representing external problems whereas, inner defected parts are not properly assessed. In recent years, research with the use of 2D and 3D MRI reconstructions on the anus levator muscle and ligament has become a hot topic. It found that the characteristic of the high resolution of soft tissue in the magnetic resonance imaging (MRI) has a big advantage in pelvic floor study.The investigators commenced the study of 3D reconstruction technology based on the MRI datasets in 2009. The investigators have mastered the most common, key technologies of MRI three-dimensional reconstruction. The investigators have done research targeted on the reconstruction methods of the normal pelvis, viscera, ligaments, pelvic floor muscles. This project is aimed at 3D reconstruction of the whole pelvic base on static and dynamic MRI images from FPOP patients, and establish the corresponding space coordinates assessment system to do location and quantitative research of the pelvic viscera and its support structure, thus providing a FPOP diagnosis platform that is more precise, direct and comprehensive.

ELIGIBILITY:
Inclusion Criteria:

1. Female who were diagnosed with pelvic organ prolapse by using Pelvic Organ Prolapse Quantification (POP-Q) exams;
2. Without history of pelvic surgery;
3. Could cooperate smoothly with valsalva maneuver.

Exclusion Criteria:

1. Combined with gynecologic malignant tumors；
2. With MRI contraindications；
3. Female who refuse to undergo MRI evaluation.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a study comparing 60 cases (POP) to 20 controls (Non POP,with normal pelvic floor support) defined by using Pelvic Organ Prolapse Quantification (POP-Q) exams.All recruits will undergo the MRI evaluation,and the basic information of them will be recorded.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-09; Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Bladder，uterus and rectum space coordinates. | september 1,2017 to september 1,2019
levator ani muscle space coordinates. | september 1,2017 to september 1,2019

SECONDARY OUTCOMES:
bladder neck, internal cervix, external cervix, anorectal junction's distance from the PCL line | september 1,2016 to september 1,2019
levator hiatus width and length, Levator symphasis gap leftside and rightside,levator plate angle. | september 1,2017 to september 1,2019
Urethral rotation Angle,posterior vesicourethral angle. | september 1,2017 to september 1,2019

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang L, Liang S, Chen C, Feng J, Chen L, Peng C, Liu P. Comparison of urethral parameters in females presenting cystoceles with and without stress urinary incontinence based on dynamic magnetic resonance imaging: are they different? Abdom Radiol (NY). 2024 Aug;49(8):2902-2912. doi: 10.1007/s00261-023-04175-7. Epub 2024 Mar 18. PMID 38498153